CLINICAL TRIAL: NCT02272725
Title: Non-steroidal Anti-inflammatory Affect on Kidneys in Endurance Distances
Acronym: NAKED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Grant S Lipman, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 31907
Record Dates: First submitted 2014-10-09; First posted 2014-10-23 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-11

CONDITIONS: Acute Kidney Injury; Exercise-associated Hyponatremia; Perceived Exertion
Keywords: ultramarathon; ibuprofen; acute kidney injury; exercise-associated hyponatremia; exertion
MeSH Terms: conditions — Acute Kidney Injury | interventions — Ibuprofen; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): tasteless and inert tablets
  Interventions: Drug: Placebo
- Ibuprofen (Active Comparator): Each tablet containing 400mg of ibuprofen
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — Ibuprofen
  Other Names: motrin
  Arms: Ibuprofen
Drug: Placebo — Tasteless and inert visually identical (to ibuprofen) pills
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The specific aim of this study is to evaluate the safety of non-steroidal anti-inflammatory drugs (NSAIDs) and their impact on renal function and/or contribution to exercise-associated hyponatremia (EAH) during an ultramarathon foot race. There is currently much debate over whether NSAID ingestion during endurance events contributes to acute kidney injury. Endurance events often ignite a "perfect storm" of physiologic insults- heat stress, dehydration, and myopathy- which can all negatively impact kidney function. There is a concern that NSAIDs may further potentiate these negative effects as well as contribute to EAH through its anti-diuretic affect. To date, no powered, prospective study has ever examined the effects of NSAIDs on either of these two biochemical outcomes

Ultramarathon endurance events, defined as any race longer than a marathon (26.2 miles), are increasing in popularity, with a 10% increase in annual participants, and more than 69,000 finishers worldwide in 2013. Considerable literature has documented alterations in serum biochemical profiles of these endurance athletes, with consistent evidence of elevated serum creatinine (Cr) levels in healthy race finishers as well as those seeking medical care. While acute renal failure in ultramarathon runners is a rare occurrence, acute kidney injury is common, ranging from 34% in a single-stage ultramarathon to 55-80% in multi-stage ultramarathons. The evidence is equivocal regarding NSAID ingestion and AKI. One study showed that runners who ingested NSAIDs prior to marathons had greater post-race creatinine levels than matched controls as well as higher rates of hospitalization and acute renal failure. However, this contrasts with several other studies that showed a marked lack of difference in creatinine levels or development of acute kidney injury between NSAID users and non-users during ultramarathons. The only randomized trial to date on this subject found no difference in serum creatinine levels between the NSAID and placebo groups at ultramarathon race end, however conclusions were limited by a small unpowered sample size.

Exercise associated hyponatremia (EAH), defined as a serum sodium concentration below 135mEq/L, is recognized as a relatively common issue in endurance running events. The incidence of EAH varies depending upon the distance of the race, with reported values of 3-28% for marathons, 23 - 38% for triathlons and 4-51% in single-stage ultramarathons. EAH is likely under-diagnosed as athletes are often asymptomatic. While EAH most often manifests as non-specific symptoms such as nausea, vomiting, dizziness, and fatigue, it can be a potentially fatal disease that can progress to encephalopathy, seizures, pulmonary edema, and death. There have been no large prospective studies examining the relationship between EAH and NSAID ingestion.

DETAILED DESCRIPTION:
This study will be conducted during the fifth stage of a 6-stage ultramarathon foot race that covers a total of 250 kilometers. Data will be collected during four separate events over the course of the coming year. All races are run by the RacingThePlanet™ 4-desert race series with locations including: Jordan, Ecuador, China, and Chile. The evening after stage 4, participants will be reminded to check in at the medical tent prior to stage 5 start, and at that time the participants will be weighed and given their study drug packet (ibuprofen or visually identical placebo). Approximately 80% of the finishers complete the 80-kilometer Stage 5 in less than 19 hours, so the majority of participants will ingest 1600mg of ibuprofen (400mg q 4 hours x 4 doses). The optimal adult dosing for analgesia is 400mg every 4 hours, with a maximum daily dose of 3200mg ((1999). Product information: Motrin™, ibuprofen. Kalamazoo, MI, Pharmacia & Upjohn Company.)

Immediately after crossing the finish line of Stage 5, participants will be reweighed, then seated in the study tent where a fingertip blood sample will be obtained via lancet and capillary collection tube (Mock, Morrison, & Yatscoff, 1995) then analyzed for Na, Cr and BUN (utilizing a Chem-8 cartridge) onsite immediately after collection using an iSTAT® point-of- care analyzer (Abbott; East Windsor, NJ). Any participant who did not complete any stage prior to stage 5 will be removed from the competition and the study. Both the point-of-care device and the digital scale will be calibrated for prior to taking measurements. At this point, the study is over and there is no further participant responsibilities.

ELIGIBILITY:
Inclusion Criteria:

* Any participant in a RacingThePlanet sanctioned event who understands the consent form in English.

Exclusion Criteria:

* Allergic to any form of non-steroidal anti-inflammatory
* Taken a NSAID or steroid in prior 12 hours
* 1 kidney
* Known to be pregnant or suspected to be pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant S Lipman, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lipman GS, Shea K, Christensen M, Phillips C, Burns P, Higbee R, Koskenoja V, Eifling K, Krabak BJ. Ibuprofen versus placebo effect on acute kidney injury in ultramarathons: a randomised controlled trial. Emerg Med J. 2017 Oct;34(10):637-642. doi: 10.1136/emermed-2016-206353. Epub 2017 Jul 5. PMID 28679502

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Ibuprofen
Started | 49 | 42
Completed | 47 | 42
Not Completed | 2 | 0
Not completed — equipment malfunction | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ibuprofen | Total
Number analyzed (Participants) | 47 | 42 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 42 | 89
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (10.5) | 40 (7.1) | 41 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 67
  Male | 13 | 9 | 22
Creatinine [Mean (Standard Deviation); unit: mg/dL] — Baseline creatinine estimated on baseline age and weight
  mg/dL | 0.83 (0.1) | 0.83 (0.1) | 0.83 (0.1)

OUTCOME MEASURES:

1. Primary Outcome: Acute Kidney Injury
Description: The participants experiencing acute kidney injury (diagnosed by an increase in creatinine of greater or equal to 1.5x that of estimated baseline creatinine from age and weight) will be from measured point-of-care blood test of the finish line immediately following the completion of a 50 mile ultramarathon. This outcome measure is a biochemical reading, that may not necessarily be a clinical adverse event.
Time Frame: participants will be followed through the duration of a 50 mile ultramarathon, an expected average of 18 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ibuprofen
Number analyzed (Participants) | 47 | 42
Participants | 16 | 22

2. Secondary Outcome: Perceived Exertion
Description: A Borg score of perceived exertion will be measured at the finish line immediately following completion of a 50 mile ultramarathon to measure what affect ibuprofen had on perceived exertion as analgesia may have made the endurance event perceived as less exertional. Scores range from 7 - 20, with higher scores indicative of greater amount of exertion.
Time Frame: participants will be followed through the duration of a 50 mile ultramarathon, an expected average of 18 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen
Number analyzed (Participants) | 47 | 42
units on a scale | 15.96 (2.6) | 15.99 (2.5)

3. Secondary Outcome: Exercise-Associated Hyponatremia
Description: The count of participants experiencing exercise-associated hyponatremia (defined as < 135 mEq) will be estimated from measured point-of-care blood test at the finish line immediately following completion of a 50 mile ultramarathon. This outcome measure is a biochemical reading, that may not necessarily be a clinical adverse event.
Time Frame: participants will be followed through the duration of a 50 mile ultramarathon, an expected average of 18 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ibuprofen
Number analyzed (Participants) | 47 | 42
Participants | 7 | 3

ADVERSE EVENTS:
Time Frame: The adverse event data was collected at the time of study completion (the finish line of the 50 mile ultramarathon) through to the finish line of the next stage of the race, approximately 24 hours.
Description: Acute renal failure as defined clinically by inability or decreased ability to make urine and / or increasing creatinine values in the 24 hours after the finish line of the ultramarathon (as checked on the basis of the runner's clinical status)
Arm/Group | Placebo | Ibuprofen
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/42
Other Adverse Events (participants affected / at risk) | 0/47 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No